CLINICAL TRIAL: NCT02157220
Title: Prospective Double-blinded Randomised Comparison of Profix Mobile to Fixed Bearing Knee Replacements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Cameron Handford, Dr Cameron Handford, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC12098
Record Dates: First submitted 2014-05-30; First posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomised group 1 (Experimental): This study is looking at a group of patients with knee osteoarthritis or other pathology requiring total knee arthroplasty. This group of patients were randomised to receive either a mobile bearing prosthesis or a fixed bearing prosthesis.
  Interventions: Device: Fixed bearing prosthesis
- Randomised group 2 (Experimental): This study is looking at a group of patients with knee osteoarthritis or other pathology requiring total knee arthroplasty. This group of patients were randomised to receive either a mobile bearing prosthesis or a fixed bearing prosthesis.
  Interventions: Device: Mobile bearing prosthesis

INTERVENTIONS:
Device: Fixed bearing prosthesis
  Arms: Randomised group 1
Device: Mobile bearing prosthesis
  Arms: Randomised group 2

SUMMARY:
This is a randomised control trial comparing two different prosthetic designs used in total knee arthroplasty. Participants were randomised to receive either of the two prostheses and then were followed up of a period of 7 years, looking at pain, range of motion and impact on quality of life. The literature and joint registry of Australia shows that one of the prosthesis may be inferior to the other. Our research team hypothesised that this was not the case and that previous elicited differences were related to other factors.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to a single orthopaedic surgeon with knee pathology, who were suitable candidates for total knee arthroplasty

Exclusion Criteria:

* refusal to participate
* other simultaneous surgery
* post traumatic osteoarthritis
* prior open knee surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-05; Primary Completion 2012-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Visual pain analogue score | 6 weeks
  Participants asked to rate their level of pain on a scale
Range of motion | 6 weeks
  The range of motion of the joint was assessed in both flexion and extension
Activities of Daily Living | 6 weeks
  Questionnaire looking at how the intervention impacts of activities of daily living
X-ray analysis of joint alignment | 5-7 year
  Using X-rays, the knee was assessed for mechanical and anatomical alignment
Visual pain analogue score | 6 months
visual pain analogue score | 12 months
visual analogue pain score | 5-7 years
range of motion | 6 months
range of motion | 1 year
range of motion | 5-7 years
activities of daily living | 6 months
activities of daily living | 1 year
activities of daily living | 5-7 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Dean Pepper, orthopaedic surgeon private rooms, Port Macquarie, New South Wales, Australia